CLINICAL TRIAL: NCT02825615
Title: Comparison of Conventional and Ultrasound Guided Techniques of Radial Artery Cannulation in Different Hemodynamic Subsets: a Randomized Controlled Study
Brief Title: Better Arterial Cannulation Technique With Different Hemodynamics
Acronym: CCURDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MREC#644
Record Dates: First submitted 2016-07-03; First posted 2016-07-07 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Acute Respiratory Failure; Shock
Keywords: radial artery cannulation; ultrasound guided; first success rate; systolic blood pressure; shock
MeSH Terms: conditions — Shock

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional method (CM) (Active Comparator): Radial artery cannulation has been done using the conventional method. Cannulation failure with this technique were tried with USG technique secondarily.
  Interventions: Procedure: Radial artery cannulation
- Ultrasound guided method (USG) (Experimental): Radial artery cannulation is done with ultrasound guidance for this group of patients. Cannulation failure with this technique were tried with Conventional technique secondarily.
  Interventions: Procedure: Radial artery cannulation

INTERVENTIONS:
Procedure: Radial artery cannulation — Radial artery cannulation done with conventional and ultrasound guidance in two respective groups of patients and their first pass success and ultimate success rates compared in different hemodynamic subsets of the patients.

SUMMARY:
Purpose Two techniques of radial artery cannulation, ultrasound guided (USG) and conventional method (CM) were compared to find the better technique in general and in different hemodynamic subsets of patients.

Method This is a prospective randomized, single center study of 100 patients. The details of the primary cannulation technique, number of attempts, time taken, failure and cross-over technique were recorded for three different hemodynamic subsets with Systolic blood pressure <80 mm hg, 80-100 mm hg and > 100 mm hg.

ELIGIBILITY:
Inclusion Criteria:

* All adult Patients worthy of radial artery cannulation, who consented

Exclusion Criteria:

* No consent

Ages: 13 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
First pass success rate | 1 year
  First pass success rate depicted the better method of cannulation of radial artery
Final/ultimate success rate of an intervention | 1 year
  If the primary technique failed then the cannulation was done with the secondary technique and hence the final success rate was calculated for each of the techniques: conventional and ultrasound guided.

SECONDARY OUTCOMES:
Time taken for the respective technique | 1 year
  Time taken for each technique was calculated from start of needle insertion till the cannula was completely inserted. The time was compared between the two arms
Attempts of cannulation | 1 year
  Number of attempts made by a technique was recorded and compared

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flumignan RL, Trevisani VF, Lopes RD, Baptista-Silva JC, Flumignan CD, Nakano LC. Ultrasound guidance for arterial (other than femoral) catheterisation in adults. Cochrane Database Syst Rev. 2021 Oct 12;10(10):CD013585. doi: 10.1002/14651858.CD013585.pub2. PMID 34637140